CLINICAL TRIAL: NCT00241007
Title: A Study Comparing Valsartan With And Without Hydrochlorothiazide In Patients With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAH631C2301E1
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2005-10

CONDITIONS: Hypertension
Keywords: HYPERTENSION, VALSARTAN
MeSH Terms: conditions — Hypertension | interventions — Valsartan

INTERVENTIONS:
Drug: VALSARTAN, VALSARTAN+HYDROCHLOROTHIAZIDE

SUMMARY:
SAFETY EXTENSION STUDY TO THE CORE STUDY CVAH631C2301

ELIGIBILITY:
Inclusion Criteria:

SUCCESSFUL COMPLETION OF STUDY CVAH631C2301

-

Exclusion Criteria:

* NONE

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 836 (Actual)
Dates: Start 2003-12; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events at each study visit for 54 weeks

SECONDARY OUTCOMES:
Change from baseline in diastolic blood pressure from baseline after 54 weeks
Change from baseline in systolic blood pressure from baseline after 54 weeks
Change from baseline in standing diastolic and systolic blood pressure after 54 weeks
Hematology and blood chemistries up to 54 weeks
Physical condition including pregnancy, pulse and weight at each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States